CLINICAL TRIAL: NCT01028690
Title: Control of Helicobacter Pylori Infection by Dietary Supplementation With Lactobacillus Reuteri
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Regional para el Estudio de las Enfermedades Digestivas (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Francisco Javier Bosques Padilla, Centro Regional Para el Estudio de las Enfermedades Digestivas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lactobacilos vs helicobacter
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Helicobacter Pylori Infection; Dyspepsia
Keywords: Helicobacter pylori; Eradication therapy; Lactobacillus reuteri; Dyspeptic symptoms
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus reuteri (Active Comparator): L. reuteri is one species of lactobacillus that naturally inhabits the gastrointestinal tract of humans
  Interventions: Dietary Supplement: Lactobacillus reuteri
- placebo (Placebo Comparator): Placebo will be delivered in a chewable tablet form (1.5g per dose)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Lactobacillus reuteri is a mixture of L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475; will be delivered at a dose of 1x108 CFU of each strain. One dose is to be taken once per day giving a dose of L. reuteri of 2x108 CFU/day. Will be taken daily throughout the entire study, from the day of inclusion to the final analysis at the end of follow-up after eradication therapy. Will be delivered either in a chewable tablet form
  Other Names: Progastria
  Arms: Lactobacillus reuteri
Dietary Supplement: Placebo — placebo
  Other Names: bioGaia
  Arms: placebo

SUMMARY:
Helicobacter pylori colonizes approximately to 50% of the world-wide population.

There is an exigency to find routes alternating to control the infection with an ample perspective but without the complications of induction of resistance to antibiotics. Supplement dietetic with Lactobacillus reuteri (L. reuteri) in humans takes to the colonization of epithelium gastric and this, combined with the observation of which L. reuteri has the capacity to inhibit the growth of H. Pylori and its union to the gastric mucosa, indicates the potential that the native human bacteria control and influence in the colonization in humans.

The acid-lactic bacteria (in particular the lactobacillus) have been studied by their effects in humans infected with H. Pylori with some success to reduce the load of bacteria Studies using supplements with L. reuteri as much in infected symptomatic patients as asymptomatic with H. pylori showed a clear reduction of the load of bacteria after 4 weeks of use and this was concordant with a reduction in the symptoms associated to the infection.

DETAILED DESCRIPTION:
The objective of this study is to determine if the dietetic supplementation with a combination of the stock of L. Reuteri (L. reuteri Progastria) is effective to control the load of bacteria and the consequences of the infection in patients infected with H. pylori.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 - 65 years
* Infection with H. pylori defined as ∆ > 20 ppm in the UBT test
* Non-ulcer dyspepsia
* No earlier eradication therapy for H. pylori infection
* Written informed consent
* Stated availability throughout the entire study period
* Mental ability to understand and willingness to fulfil all the details of the protocol

Exclusion Criteria:

* Duodenal or gastric ulcer
* MALT lymphoma
* Penicillin allergy
* Gastric resection (at any time)
* First level relatives of gastric cancer patients
* Absence of GI symptoms
* Use of NSAIDs, aspirin or other anti-inflammatory drugs within 1 week (for occasional use) or 3 weeks (for chronic use) of inclusion
* Use of oral antibiotics and/or PPIs and/or H2-antagonists during the 2 weeks prior to ingestion of the study product
* Pregnancy
* Participation in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-09 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Assessed decrease H. pylori gastric load by histology after 28 days compared to placebo and assessed by 13C-UBT before and after 28 days use of L. compared to placebo | 28 days

SECONDARY OUTCOMES:
To decrease dyspeptic symptoms before, during and after eradication therapy as assessed by a gastro-intestinal symptom rating scoring within and between L. reuteri and placebo-supplemented subjects | 101 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Bosques, MD PhD, Principal Investigator — Centro Regional para el Estudio de las Enfermedades Digestivas
Locations (1):
- Centro Regional para el Estudio de las Enfermedades Digestivas, Facultad de Medicina y Hospital Universitario, UANL, Monterrey, Nuevo León, Mexico